CLINICAL TRIAL: NCT04179058
Title: Interstitial Pneumonia With Autoimmune Features: Evaluation of Connective Tissue Disease Incidence During Follow-up
Acronym: EVOLIPAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI251
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Idiopathic Interstitial Pneumonia
Keywords: Connective tissue disease; Interstitial lung disease; Interstitial pneumonia with autoimmune features
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias; Connective Tissue Diseases; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPAF patients: IPAF definition according to 2015 ERS/ATS criteria
  Interventions: Other: Follow-up
- non-IPAF patients
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Clinical data, radiological data and laboratory tests follow-up

SUMMARY:
Interstitial lung diseases (ILD) represent a frequent complication of connective tissue diseases (CTDs), especially systemic sclerosis, idiopathic inflammatory myopathies and rheumatoid arthritis. ILD can either occur during CTD course or be the first manifestation of CTDs. Therefore screening patients with ILD for CTD is crucial. In some cases, ILD are associated with clinical and/or serological autoimmune features but not classifiable for CTDs. Evolution of these forms to defined CTDs has never been study. Recently, the European Respiratory Society/American Thoracic Society experts proposed a new term, "interstitial pneumonia with autoimmune features" or IPAF, to describe these patients according to updated classification criteria. Aims of this study were to compare CTD occurence during follow-up between IPAF and non-IPAF patients in a idiopathic interstitial pneumonia cohort and to identify risk factors of CTD progression in IPAF patients at diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of ILD confirmed by two chest-HRCT 3 months apart
* Patients with a minimal follow-up duration of 3 years after ILD diagnosis

Exclusion Criteria:

* Patients with a defined CTD at ILD diagnosis
* Patients with an other ILD etiology identified at diagnosis (i.e. sarcoidosis, hypersensitivity pneumonitis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic interstitial pneumonia classifiable or not as IPAF
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
CTD incidence | After 3 years of follow-up
  CTD incidence according to classification criteria: rheumatoid arthritis (2010 ACR/EULAR criteria), systemic erythematosus lupus (2019 ACR/EULAR criteria), Sjögren syndrome (2016 ACR/EULAR criteria), systemic sclerosis (2013 ACR/EULAR criteria), idiopathic inflammatory myopathies (2017 ACR/EULAR criteria) and mixed connective tissue disease (modified Sharp criteria or Alarcon-Segovia criteria or Kasukawa criteria)

SECONDARY OUTCOMES:
IPAF clinical domain criteria | Baseline
  "mechanic hands", Gottron's sign, distal digital tip ulceration, inflammatory arthritis or polyarticular joint stiffness > 60mn, telangiectasia, Raynaud's phenomenon, unexplained digital oedema
IPAF serological domain criteria | Baseline
  ANA titre and pattern, RF, anti-CCP, anti-dsDNA, anti-Ro, anti-La, anti-ribonucleoprotein, anti-Smith, anti-Scl70, anti-tRNA synthetase, anti-PM-Scl, anti-MDA5
IPAF morphological domain criteria | Baseline
  NSIP, and/or OP, or LIP radiology pattern by HRCT
ILD severity | Baseline, 6 months of follow-up and at the last visit
  PFT (pulmonary function test): FVC, FEV1, DLCO (percentages of predicted values)
Survival rate | After 3 years and 5 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roland JAUSSAUD, Pr, Principal Investigator — Central Hospital, Nancy, France
Locations (2):
- France (2):
  - Central Hospital, Lille
  - Central Hospital, Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steen VD, Medsger TA. Changes in causes of death in systemic sclerosis, 1972-2002. Ann Rheum Dis. 2007 Jul;66(7):940-4. doi: 10.1136/ard.2006.066068. Epub 2007 Feb 28. PMID 17329309
- [Background] Fathi M, Dastmalchi M, Rasmussen E, Lundberg IE, Tornling G. Interstitial lung disease, a common manifestation of newly diagnosed polymyositis and dermatomyositis. Ann Rheum Dis. 2004 Mar;63(3):297-301. doi: 10.1136/ard.2003.006122. PMID 14962966
- [Background] Tanaka N, Kim JS, Newell JD, Brown KK, Cool CD, Meehan R, Emoto T, Matsumoto T, Lynch DA. Rheumatoid arthritis-related lung diseases: CT findings. Radiology. 2004 Jul;232(1):81-91. doi: 10.1148/radiol.2321030174. Epub 2004 May 27. PMID 15166329
- [Background] Keane MP, Lynch JP 3rd. Pleuropulmonary manifestations of systemic lupus erythematosus. Thorax. 2000 Feb;55(2):159-66. doi: 10.1136/thorax.55.2.159. No abstract available. PMID 10639536
- [Background] Tillie-Leblond I, Wislez M, Valeyre D, Crestani B, Rabbat A, Israel-Biet D, Humbert M, Couderc LJ, Wallaert B, Cadranel J. Interstitial lung disease and anti-Jo-1 antibodies: difference between acute and gradual onset. Thorax. 2008 Jan;63(1):53-9. doi: 10.1136/thx.2006.069237. Epub 2007 Jun 8. PMID 17557770
- [Background] Kinder BW, Collard HR, Koth L, Daikh DI, Wolters PJ, Elicker B, Jones KD, King TE Jr. Idiopathic nonspecific interstitial pneumonia: lung manifestation of undifferentiated connective tissue disease? Am J Respir Crit Care Med. 2007 Oct 1;176(7):691-7. doi: 10.1164/rccm.200702-220OC. Epub 2007 Jun 7. PMID 17556720
- [Background] Vij R, Noth I, Strek ME. Autoimmune-featured interstitial lung disease: a distinct entity. Chest. 2011 Nov;140(5):1292-1299. doi: 10.1378/chest.10-2662. Epub 2011 May 12. PMID 21565966
- [Background] Fischer A, West SG, Swigris JJ, Brown KK, du Bois RM. Connective tissue disease-associated interstitial lung disease: a call for clarification. Chest. 2010 Aug;138(2):251-6. doi: 10.1378/chest.10-0194. PMID 20682528
- [Background] Fischer A, Antoniou KM, Brown KK, Cadranel J, Corte TJ, du Bois RM, Lee JS, Leslie KO, Lynch DA, Matteson EL, Mosca M, Noth I, Richeldi L, Strek ME, Swigris JJ, Wells AU, West SG, Collard HR, Cottin V; "ERS/ATS Task Force on Undifferentiated Forms of CTD-ILD". An official European Respiratory Society/American Thoracic Society research statement: interstitial pneumonia with autoimmune features. Eur Respir J. 2015 Oct;46(4):976-87. doi: 10.1183/13993003.00150-2015. Epub 2015 Jul 9. PMID 26160873